CLINICAL TRIAL: NCT03130647
Title: The Effects of Transcranial Focused Ultrasound on Human Motor Learning
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Left university
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M1 ultrasound
Record Dates: First submitted 2017-03-16; First posted 2017-04-26 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Repeated measures sham controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Focused ultrasound (Experimental): Repeated measures sham control
  Interventions: Device: Focused ultrasound

INTERVENTIONS:
Device: Focused ultrasound — Focused ultrasound

SUMMARY:
Transcranial focused ultrasound (tFUS) is a form of neuromodulation that uses a single element transducer to produce highly focused low-intensity acoustic energy that can be used to affect cortical excitability in humans.

DETAILED DESCRIPTION:
Here the investigator plan to investigate the effect of tFUS on motor behavior. M1 has been chosen for two fundamental reasons for this study: 1) The use of muscle contraction to generate a detectable evoked potential signal allows for targeting of a precise area within M1 with tFUS, and 2) It is known that M1 is involved in fast learning of sequential motor tasks By targeting M1 with tFUS in neurologically healthy volunteers, we can study the effects of tFUS on motor learning measures (e.g., reaction time, accuracy) while a subject is performing a finger tapping motor learning task. If ultrasound is proven efficacious for stimulating the motor cortex, non-surgical ultrasound could potentially replace costly and risky surgery for the treatment of brain disorders as is common with deep brain stimulation for essential tremor or Parkinson's disease. There is currently no way to affect brain tissue deep into the cortex without surgery, genetic alteration or viral vectors (the latter two are not approved for human use). This technology is non-surgical and as invasive as any diagnostic ultrasound exam. With success, transcranial focused ultrasound could become useful world-wide as a cheap, portable and effective tool for human brain mapping efforts as well as for the diagnosis and potential treatment of a broad range of psychiatric and neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age Provide written informed consent

Exclusion Criteria:

* Evidence of a current significant medical illness or psychiatric or central or peripheral neurologic disorder History of loss of consciousness of more than ten minutes in the past year or loss of consciousness in a lifetime that required rehabilitation services Personal or family history of seizure Any history of stroke/transient ischemic attack (TIA) Taking any medications that may decrease the threshold for seizure Pregnancy Affirmative answers to one or more questions of the provided attached safety questionnaires. These are not absolute contraindications to this study but the risk/benefit ratio will be carefully balanced by the PI Left handedness. Failure to follow laboratory or study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
Reaction Time | 4 months
  Reaction time to visual stimulus response task

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No sharing plan